CLINICAL TRIAL: NCT05073341
Title: Effectiveness of Nurse-led Family Intervention on Stress, Engagement With Patient's Care and Satisfaction Among Primary Caregivers of Chronic Liver Disease Patients Admitted in High Dependency Unit of ILBS, New Delhi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ILBS-CLD-01
Record Dates: First submitted 2021-10-08; First posted 2021-10-11 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2021-10

CONDITIONS: Family Members of the Patients

STUDY DESIGN:
Intervention Model Description: Quasi experimental design
Masking Description: non randomisation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental and control group and intervention is given in the experimental group (Experimental): Nurse-led family intervention is given in the experimental group having three components i.e infarmation about the patient condition , guidance, and emotional support
  Interventions: Other: Nurse-led family intervention
- control group (Other): No intervention will be given in the control group
  Interventions: Other: Nurse-led family intervention

INTERVENTIONS:
Other: Nurse-led family intervention — Nurse-led family intervention having three components first is infarmation about the patient's condition and guidance will be given to solve there queries and the emotional support will be given to the primary caregivers of CLD patient's admitted in HDU

SUMMARY:
Quasi experimental study to check the effectiveness of Nurse-led family Intervention on stress, engagement with patient care and satisfaction among primary caregivers of chronic liver disease patients admitted in high depency unit ILBS, two group pre test post test design non randomisation with the Nurse-led family intervention with the sample size of 80 using purposive sampling technique and having independent variable as Nurse-led family intervention and dependent variables are stress, Engagement with patient care and satisfaction and these variables are assesed by using kingston caregivers scale(KCSS) caregiver health engagement scale (CHEW-S)and one knowledge questionnaire based on engagement and satisfaction scale

DETAILED DESCRIPTION:
study having different inclusion and exclusion for criteria CLD patients and Caregiver sof patint's admitted in HDU inclusion criteria of primary caregivers between the age group of 18-65years understand hindi and english duration of hjospitalization should be more than 6 hours exclusion criteria is primary are givers who cannot understand hindi or english and age more than 65 years of age , craegivers of patients who are having disease other than CLD and those who are not willing to participate inclusion for criteria CLD patients decompensated CLD patients , understand hindi and english , duration of hospitalization more than 6 hours , patient is concious and in semi concious state and patient with hepatic encephlopathy

ELIGIBILITY:
Inclusion Criteria:between age group of 18-65 years

* primary caregivers of CLD patient's understand hindi and english duration of hospitalization more than 6 hours

Exclusion Criteria:

* primary caregivers who cannot understand hindi and english age more than 65 years of age caregivers of patient's who are other than CLD not willing to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
to reduce stress, increase satisfaction and increse the engagement with patient care | one month data collection
  stress will be reduced by giving guidance and emotional support and infarmation about their patient condition

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No